CLINICAL TRIAL: NCT01310621
Title: Surfactant Lung Lavage Versus Standard Care In The Treatment Of Meconium Aspiration Syndrome- A Randomized Controlled Study
Brief Title: Comparison Of Surfactant Lung Lavage With Standard Care In The Treatment Of Meconium Aspiration Syndrome
Acronym: Sur-Lu-Lav
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, Sushma Nangia, M.D., Professor of Pediatrics, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LHMC/2011/Sur-Lu-Lav
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Meconium Aspiration Syndrome
Keywords: Neonate; Meconium aspiration syndrome; surfactant lung lavage
MeSH Terms: conditions — Meconium Aspiration Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Lavage (No Intervention): Neonate randomized to this group will be managed as per the standard protocol in the neonatal ward. The evaluation of respiratory distress will be done using Downe's score at hourly intervals till 24 hrs, followed by 2 hourly intervals till 72 hrs and finally 4 hourly intervals till resolution of clinical distress.
- Surfactant Lavage (Experimental): The diluted surfactant is instilled into endotracheal tube over a period of 15 to 20 seconds. Once the instillation is complete, 5 manual breaths will be provided and infant will be repositioned supine. The suction catheter will be inserted and advanced to a position approximately 5mm past the end of endotracheal tube. Suction will be activated for no more than 10 seconds and would be temporarily halted earlier if the oxygen saturation value falls by > 5% of the prelavage value. The same shall be resumed once prelavage oxygen saturation has been restored. The infant's bed will now be moved back to horizontal position. Once the neonate is STABLE, suctioning will be again repeated. The total retrieved volume is measured and recorded.This procedure will be done in both right and left lateral decubitus position
  Interventions: Drug: Bovine surfactant

INTERVENTIONS:
Drug: Bovine surfactant — * Dose of diluted surfactant : 20ml/kg
  * Type :Bovine surfactant
  * Phospholipid concentration: 5 mg/ml
  * Number of lavages to be given: 2 (10ml/kg each)
  Arms: Surfactant Lavage

SUMMARY:
The purpose of this study is to evaluate the role of surfactant lung lavage in the treatment of meconium aspiration syndrome. Aspiration of meconium into the tracheo-bronchial tree with the onset of respiration results in meconium aspiration syndrome (MAS). Aspirated meconium inhibits surfactant function directly and also decreases its synthesis by its toxic effects on type 2 pneumocytes. There is no specific treatment recommended for meconium aspiration syndrome. Numerous studies have shown that exogenous surfactant improves outcome in babies with meconium aspiration. Surfactant replacement alone does not remove meconium from airways and multiple doses may be required .Therefore an effective therapy to improve outcome is crucial in treating infants with meconium aspiration. Surfactant Lung lavage has been shown to be alternative to bolus therapy in treating neonates with meconium aspiration as shown by many pilot studies. So the investigators have decided to study the role surfactant lung lavage in the treatment of meconium aspiration syndrome.

DETAILED DESCRIPTION:
Meconium is an odourless, thick, blackish green material first demonstrable in the foetal intestinal tract during the third month of gestation. Approximately 10-15% of deliveries are complicated by the passage of meconium around the time of delivery. The risk of meconium stained amniotic fluid (MSAF) is strongly correlated with gestational age. An adverse intrauterine environment with resultant foetal asphyxia is proposed as the most common explanation for MSAF.

Aspiration of meconium into the tracheo-bronchial tree with the onset of respiration results in meconium aspiration syndrome (MAS). MAS is defined as respiratory distress with compatible chest x-ray finding in an infant born through MSAF whose symptoms cannot be otherwise explained. Despite current interventions such as intubation with tracheal suction, it is estimated that 5-20 % of infants born through MSAF develop MAS. It represents a leading cause of perinatal morbidity. Approximately 50% of the infants with MAS require mechanical ventilation; 15%-30% develop pulmonary air leaks and 5%-12% die.

The pathophysiology of meconium aspiration syndrome includes airway obstruction, surfactant inactivation, inflammation and pulmonary hypertension. Meconium itself inactivates the surfactant in the alveoli and its presence also causes secondary surfactant deficiency as meconium is toxic to type 2 alveolar cells which secrete surfactant. There is no specific treatment recommended for meconium aspiration syndrome .Treatment for MAS is generally supportive and includes supplemental oxygen as needed, assisted ventilation to maintain lung volume and improve gas exchange, and circulatory support with volume resuscitation and vasopressor infusions to maintain adequate perfusion. Successful treatment of meconium aspiration relies on effective meconium removal without inactivating or washing out surfactant, followed by appropriate ventilator care.

Surfactant replacement in neonates with severe meconium aspiration syndrome has been shown to improve oxygenation and reduce the severity of respiratory failure, air leaks and need for extracorporeal membrane oxygenation.

Surfactant replacement alone does not remove the meconium present in the airways and hence multiple doses may be required. Therefore an effective strategy to improve outcome in neonates with MAS needs to not only remove meconium but also retain the surfactant for adequate lung expansion and function.

Lung lavage using diluted surfactant has recently been shown to be an alternative to bolus therapy in treating MAS. This has advantage of removing surfactant inhibitors from alveolar space, in addition to augmenting surfactant concentration in alveolar space. Initial pilot case series using surfactant lung lavage have shown promise and there is a need to systematically study this in a RCT. The same has also been expressed in the literature on this subject. Hence the purpose of this prospective randomized controlled trial is to compare the efficacy of surfactant lung lavage over standard therapy in the treatment of meconium aspiration syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Gestation age ≥ 37 week
* Cephalic presentation
* Singleton pregnancy
* Presence of meconium stained amniotic fluid or staining of meconium in skin,umbilical cord or nails.
* Non vigorous babies
* Presence of respiratory distress(Downes score ≥4)
* Presence of meconium below vocal cords or chest x ray suggestive of meconium aspiration
* Age < 2 hours

Exclusion Criteria:

* Major congenital malformations
* Congenital heart disease
* Hydrops fetalis
* Air leaks
* Pulmonary hemorrhage

Ages: 30 Minutes to 2 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
duration of oxygen therapy in hours | till discharge or death
  The duration of oxygen therapy, mode of delivery, FiO2 and flow rate will be documented hourly within first 2 hours before lavage and in post lavage- hourly up to first 24 hours, 2 hourly up to 72 hours and 4 hourly thereafter till the cessation of oxygen therapy
Severity of respiratory distress | till discharge or death
  The severity of respiratory distress will be assessed using Downe's Score. These parameters will be documented hourly within first 2 hours before lavage and in post lavage hourly up to first 24 hours, 2 hourly up to 72 hours and 4 hourly thereafter till the cessation of respiratory distress
need for mechanical ventilation | till discharge or death
  The babies will be assessed for the need for mechanical ventilation as per standard unit protocols.

SECONDARY OUTCOMES:
Duration of mechanical ventilation | till discharge or death
  Total duration of mechanical ventilation, mode and ventilator parameters are noted till the baby is on mechanical ventilation.
Complications | till discharge
  Incidence of PPHN by Echocardiography and Pneumothorax by transillumination confirmed by chest x-ray.
Incidence of sepsis | till discharge
  Incidence of sepsis defined as -
  1. SUSPECTED SEPSIS - Sepsis Screen > 2 parameters positive and/or
  2. CONFIRMED SEPSIS - Sepsis Screen positive + Blood or CSF culture positive for bacteria.
  Sepsis Screen
  1. Total leukocyte count < 5000/mm3
  2. Absolute neutrophil count < 1800/cu.mm.(Low counts as per Manroe chart for term neonates)
  3. Immature/total neutrophil ratio > 0.2
  4. Micro-ESR > 15mm in 1st hour
  5. C Reactive Protein (CRP) > 1 mg/dl
Mortality | till discharge
Duration of Hospital stay | till discharge

CONTACTS AND LOCATIONS:
Overall Officials: Sushma Nangia, MBBS, MD, DM, Study Chair — Lady Hardinge Medical College, New Delhi, India
Locations (1):
- Kalawati Saran children's Hospital, Lady Hardinge Medical College, New Delhi, National Capital Territory of Delhi, India